CLINICAL TRIAL: NCT05428150
Title: Randomized, Crossover, Multi-Dose, Steady State, Comparative Pharmacokinetics and Relative Bioavailability Study of EXCL-100 Pirfenidone-Sustained Release Tablet (EXCL-100), and Esbriet® in Healthy Volunteers
Brief Title: Randomized, Crossover, Multi-Dose Pharmacokinetics of EXCL-100 Pirfenidone-Sustained Release Tablet and Esbriet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Excalibur Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EXCL-100-102
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (Active Comparator): Esbriet® 801 mg (267 mg oral capsule x 3), three times daily (TID) with meals (6 hours apart) for 3 days, total daily dose of 2403 mg, given under fed conditions. Subjects will receive a single dose on Day 4 after breakfast.
  Interventions: Drug: Esbriet 267 MG Oral Capsule
- Regimen B (Experimental): EXCL-100, 1200 mg (600 mg oral tablet x 2), twice daily with meals (BID, every 12 hours) for 3 days, total daily dose of 2400 mg, given under fed conditions. Subjects will receive a single dose on Day 4 after breakfast.
  Interventions: Drug: EXCL-100, 600 MG Oral Tablet

INTERVENTIONS:
Drug: Esbriet 267 MG Oral Capsule — Reference Formulation
  Arms: Regimen A
Drug: EXCL-100, 600 MG Oral Tablet — Test Formulation
  Arms: Regimen B

SUMMARY:
This is a randomized, open-label, 2-treatment, 2-period, crossover steady state study conducted to evaluate the comparative bioavailability/bioequivalence of pirfenidone after multi-dose administration of EXCL-100 at doses of 1200 mg (600 mg x 2) in the fed state, and Esbriet® 801 mg (267 mg capsule x 3) given in the fed state, to healthy volunteers.

DETAILED DESCRIPTION:
After signing the Institutional Review Board (IRB) approved Informed Consent Form (ICF), subjects will undergo a screening evaluation up to 28 days prior to dosing on Day 1 of Period 1. Subjects who satisfy the screening evaluation and who meet the inclusion and exclusion criteria will be enrolled in the study. Subjects will receive multiple doses of study drug according to their assigned sequence of treatment in Period 1. After completion of study procedures, a washout period will be completed prior to crossover to Period 2 to receive the second treatment in their sequence. Subjects will receive Regimens A (Esbriet® 801 mg three times daily with meals for 3 days) and B (EXCL-100, 1200 mg twice daily with meals) according to the randomization schedule. Pharmacokinetic (PK) blood samples will be taken on multiple days during the study periods.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female aged 18 to 65 years inclusive with a body mass index at time of screening between 18 and 32 kg/m2.
2. Subject is in good health, as determined by the investigator, as documented by the medical history, physical examination, vital sign assessment, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and general observations.

   1. Abnormalities or deviations outside the normal ranges for any clinical assessments (laboratory tests, ECG, vital signs) may be repeated once during the screening period at the discretion of the Investigator(s), and results that continue to be outside the normal ranges must be judged by the investigator to be not clinically significant and acceptable for study participation.
   2. At Screening, ALT, AST, and total bilirubin values must be ≤ 1.5 times the upper limit of normal (ULN).
   3. All other laboratory test results that are outside the normal range at Screening and judged by the investigator to be not clinically significant, may be repeated. Results that continue to be outside the normal range must be judged by the investigator to be not clinically significant and acceptable for study participation.
3. Male and female

   1. Female subjects of childbearing potential who are not pregnant as confirmed by a negative serum pregnancy test at Screening and urine pregnancy test on Day -1 of Period 1, non-lactating, using effective methods of contraception for a minimum of one complete menstrual cycle prior to the Screening visit and agree to continue using until 30 days after the last dose of study drug. Effective methods of birth control include: Hormonal methods of contraception including oral contraceptives containing combined estrogen and progesterone, a vaginal ring, injectable and implantable hormonal contraceptives, intrauterine hormone-releasing system (eg, Mirena) and progestogen-only hormonal contraception associated with inhibition of ovulation, nonhormonal intrauterine device (IUD), bilateral tubal occlusion, or vasectomized partner, if that partner is the sole sexual partner.
   2. Female subjects of non-childbearing potential must be surgically sterile (e.g., hysterectomy, bilateral tubal ligation, bilateral salphingectomy and/or bilateral oophorectomy) or post-menopausal (no menses for >1 year with follicle stimulating hormone [FSH] in the post-menopausal range at screening, based on the central laboratory's range).
   3. Female subject must not donate eggs during the study and for at least 30 days after the last dose of study drug.
   4. Male subjects who have not had a vasectomy must agree to use an effective method of contraception (condom with spermicide) during the study and until 90 days after the last dose of the study drug, and to not donate sperm during the study and for at least 90 days after the last dose of study drug.
4. Subject is willing to remain in the study facility for the duration of the confinement periods.
5. Subject is able to communicate with the investigator and is willing to comply with the requirements of the entire study.
6. Subject understands and signs the informed consent form.

Exclusion Criteria:

1. History or presence of clinically significant (CS) cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, psychiatric, or other major disease, as determined by the Investigator.
2. Any surgical or medical condition that could interfere with the absorption, distribution, metabolism, or excretion of the drug.
3. History of severe allergic or anaphylactic reactions.
4. Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C virus antibody (HCV), or positive human immunodeficiency virus (HIV) test result at Screening.
5. A positive result on SARS-CoV-2 (COVID-19) tests assessed by rapid antigen testing (RAT) at Day -1 of Period 1.
6. History of alcohol abuse or illicit drug use within 1 year of Screening or consumption of alcohol greater than 21 units per week. A unit of alcohol is equivalent to 1 can of beer, 1 glass of wine, or the equivalent of 1 alcoholic drink.
7. A positive urine drug or breath alcohol test result at Screening or Day -1 of Period 1.
8. Smoking and the use of nicotine-containing products (including nicotine patches, gum, inhalers, and e-cigarettes) within 6 months of the Screening visit or positive urine cotinine tests at Screening or Day -1 of Period 1) and inability to refrain from nicotine from Screening until the end of the study.
9. Standard donation of blood or blood products within 30 days of Day-1 of Period 1 .
10. Use of any investigational drug within 30 days of Day-1 of Period 1 .
11. Participants previously dosed in any pirfenidone clinical study.
12. Use of CYP1A2 inhibitors (e.g., enoxacin, ciprofloxacin) or CYP1A2 inducers within 14 days prior to screening and for the duration of the study.
13. Participants who have received fluvoxamine therapy within 28 days before screening.
14. Need for concomitant prescription medications, except for birth control and hormone replacement therapy, starting 14 days or 5 half-lives before dosing (Day 1 of Period 1), whichever is longer, through the completion of all study procedures, or subject needs an over the counter (OTC) medication including other herbal supplements or multivitamins, starting 7 days before dosing (Day 1 of Period 1) through the completion of all study procedures. Up to 2 grams per day of acetaminophen is allowed at the discretion of the PI.
15. Regular caffeine consumption of greater than 300 mg/day. Inability to restrict consumption of caffeine to less than 300 mg/day (2 standard cups brewed coffee) during the study.
16. Seated blood pressure was less than 90/40 mmHg or greater than 140/90 mmHg at screening. (After being seated for at least 5 minutes). Measurements can be repeated once to determine eligibility.
17. Heart rate was less than 40 bpm or great than 99 bpm at screening. (After being seated for at least 5 minutes). Measurements can be repeated once to determine eligibility.
18. Participants with calculated creatinine clearance rate less than (<) 60 milliliters per min (mL/min) (calculated using the CKD-EPI equation) at screening.
19. Any clinically significant ECG abnormality at screening (as deemed by the Investigator and the Sponsor's Medical Monitor).
20. QTcF interval > 450 msec (the average value for the triplicate ECG at Screening and Day -1 of Period 1), or history of prolonged QT syndrome.
21. Other unspecified reasons that, in the opinion of the PI or Sponsor, make the subject unsuitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
AUC 0-inf | Up to Day 6 of Periods 1 and 2
  Area under plasma concentration-time curve from time 0 to infinity for pirfenidone and 5-carboxy pirfenidone

SECONDARY OUTCOMES:
AUC 0-24ss | Day 3 of Periods 1 and 2
  Area under plasma concentration-time curve from time 0 to 24 hours for pirfenidone and 5-carboxy pirfenidone
AUC last | Up to Day 6 of Periods 1 and 2
  Time 0 to the time of the last quantifiable plasma concentration for pirfenidone and 5-carboxy pirfenidone
C max | Up to Day 6 of Periods 1 and 2
  Observed maximum concentration for pirfenidone and 5-carboxy pirfenidone
Safety and Tolerability | From Day 1 of Period 1 through study completion (an average of 15 days)
  Adverse Events reported

CONTACTS AND LOCATIONS:
Overall Officials: Renu Gupta, MD, Study Director — Chief Medical Officer
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided